CLINICAL TRIAL: NCT02139644
Title: A 12-Week, Double-Blind, Placebo-Controlled, Efficacy and Safety Study of Fluticasone Propionate Multidose Dry Powder Inhaler Compared With Fluticasone/Salmeterol Multidose Dry Powder Inhaler in Adolescent and Adult Patients With Persistent Asthma Symptomatic Despite Low-dose or or Mid-dose Inhaled Corticosteroid Therapy
Brief Title: Study of Fluticasone Propionate MDPI Compared With Fluticasone/Salmeterol MDPI in Adolescent and Adult Patients With Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FSS-AS-301; 2014-001149-25 (EudraCT Number)
Record Dates: First submitted 2014-05-09; First posted 2014-05-15 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Asthma
Keywords: fluticasone propionate; multidose dry powder inhaler
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Salmeterol Xinafoate; Albuterol; Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- FS MDPI 100 / 12.5 mcg (Experimental): Patients took 1 inhalation using a multidose dry powder inhaler (MDPI) twice a day of fluticasone propionate 100 mcg (for a total daily dose of 200 mcg) and salmeterol 12.5 mcg (for a total daily dose of 25 mcg) for 12 weeks.
  Albuterol/salbutamol hydrofluoroalkane (HFA) metered dose inhaler (MDI) was supplied to participants throughout the study to be used as needed as a rescue medication.
  Interventions: Drug: FS MDPI; Drug: albuterol/salbutamol; Drug: Beclomethasone dipropionate
- FS MDPI 50 / 12.5 mcg (Experimental): Patients took 1 inhalation using a multidose dry powder inhaler (MDPI) twice a day of fluticasone propionate 50 mcg (for a total daily dose of 100 mcg) and salmeterol 12.5 mcg (for a total daily dose of 25 mcg) for 12 weeks.
  Albuterol/salbutamol hydrofluoroalkane (HFA) metered dose inhaler (MDI) was supplied to participants throughout the study to be used as needed as a rescue medication.
  Interventions: Drug: FS MDPI; Drug: albuterol/salbutamol; Drug: Beclomethasone dipropionate
- Fp MDPI 100 mcg (Experimental): Patients took 1 inhalation using a multidose dry powder inhaler (MDPI) twice a day of fluticasone propionate 100 mcg for a total daily dose of 200 mcg for 12 weeks.
  Albuterol/salbutamol hydrofluoroalkane (HFA) metered dose inhaler (MDI) was supplied to participants throughout the study to be used as needed as a rescue medication.
  Interventions: Drug: Fp MDPI; Drug: albuterol/salbutamol; Drug: Beclomethasone dipropionate
- Fp MDPI 50 mcg (Experimental): Patients took 1 inhalation using a multidose dry powder inhaler (MDPI) twice a day of fluticasone propionate 50 mcg for a total daily dose of 100 mcg for 12 weeks.
  Albuterol/salbutamol hydrofluoroalkane (HFA) metered dose inhaler (MDI) was supplied to participants throughout the study to be used as needed as a rescue medication.
  Interventions: Drug: Fp MDPI; Drug: albuterol/salbutamol; Drug: Beclomethasone dipropionate
- Placebo MDPI (Placebo Comparator): The placebo multidose dry powder inhaler was identical to the devices used to deliver active drug, and indistinguishable from the active treatments. Patients took one inhalation twice a day (approximately 12 hours apart).
  Albuterol/salbutamol hydrofluoroalkane (HFA) metered dose inhaler (MDI) was supplied to participants throughout the study to be used as needed as a rescue medication.
  Interventions: Drug: Placebo MDPI; Drug: albuterol/salbutamol; Drug: Beclomethasone dipropionate

INTERVENTIONS:
Drug: FS MDPI — FS MDPI is an inhalation-driven multidose dry powder inhaler (MDPI) containing fluticasone propionate (Fp) and salmeterol xinafoate (Sx) dispersed in a lactose monohydrate excipient and contained within a reservoir. A metered dose of drug is delivered to a dose cup via an air pulse activated when the cap is opened.
  During the treatment period, participants were randomized to either 100/12.5 mcg Fp/Sx or 50/12.5 mcg Fp/Sx in the morning and evening for a total daily dose of 200/25 mcg or 100/25 mcg Fp/Sx.
  Participants were instructed to rinse their mouth and expectorate (not swallow) after study drug administration.
  Other Names: fluticasone propionate; inhaled corticosteroid; salmeterol xinafoate; β2 adrenoceptor agonist
  Arms: FS MDPI 100 / 12.5 mcg; FS MDPI 50 / 12.5 mcg
Drug: Fp MDPI — Fp MDPI is an inhalation-driven multidose dry powder inhaler (MDPI) containing fluticasone propionate dispersed in a lactose monohydrate excipient and contained within a reservoir. A metered dose of drug is delivered to a dose cup via an air pulse activated when the cap is opened.
  During the treatment period, participants were randomized to either 100 mcg or 50 mcg of Fp one inhalation twice a day for a total daily dose of 200 mcg or 100 mcg.
  Participants were instructed to rinse their mouth and expectorate (not swallow) after study drug administration.
  Other Names: fluticasone propionate; inhaled corticosteroid
  Arms: Fp MDPI 100 mcg; Fp MDPI 50 mcg
Drug: Placebo MDPI — Placebo administered via a multidose dry powder inhaler (MDPI) one puff in the morning and one puff in the evening for 12 weeks.
  Other Names: inert powder
  Arms: Placebo MDPI
Drug: albuterol/salbutamol — A short-acting β2-adrenergic agonists (SABA), albuterol/salbutamol hydrofluoroalkane (HFA) metered dose inhaler (MDI), was provided to be used as needed for the relief of asthma symptoms during both the run-in and treatment periods (to replace the subject's current rescue medication).
  Other Names: short-acting β2-adrenergic agonists
Drug: Beclomethasone dipropionate — QVAR (beclomethasone dipropionate) 40 mcg inhalation aerosol is a pressurized MDI that contains a Food and Drug Administration (FDA)-approved formulation of beclomethasone dipropionate. Patients took 1 puff twice a day from open-label QVAR 40 mcg hydrofluoroalkane (specifically, HFA-134a) metered-dose inhaler (MDI) for the duration of the Run-in Period (14-21 days) and prior to randomization. A clinically equivalent dose of inhaled corticosteroid (ICS) was substituted in countries where QVAR 40 mcg was not available.
  Other Names: QVAR

SUMMARY:
The primary objective of this study was to evaluate the efficacy of fluticasone propionate multidose dry powder inhaler (Fp MDPI) and fluticasone propionate/salmeterol xinafoate multidose dry powder inhaler (FS MDPI) when administered over 12 weeks in patients 12 years of age and older with persistent asthma.

Study drug and placebo was supplied in Teva multidose dry powder inhaler (MDPI) devices and provided for participants to use at home. Participants performed spirometry at every visit. Each participant was given a diary at each visit for use until the next visit. Rescue medication (albuterol/salbutamol) was dispensed at each visit, if needed, as determined by the investigational center personnel.

ELIGIBILITY:
Inclusion Criteria:

1. Best pre-bronchodilator forced expiratory volume in 1 second (FEV1) of 40 to 85% of their predicted normal value.
2. Current Asthma Therapy: Patients must have a short-acting β2-agonist (for rescue use) for a minimum of 8 weeks before the Screening Visit (SV) and a low-dose inhaled corticosteroid (ICS). The low-dose ICS may be either as ICS monotherapy or as an ICS/long-acting beta agonist (LABA) combination. The ICS component of the patient's asthma therapy should be stable for a minimum of 1 months before providing consent.
3. Reversibility of Disease: Patients must have at least 15% reversibility (all patients) and at least a 200 mL increase from baseline FEV1 (patients age 18 and older) within 30 minutes after 2 to 4 inhalations of albuterol/salbutamol at the SV. Note: Patients who do not qualify for the study due to failure to meet reversibility will be permitted to perform a retest once within 7 days.
4. Patients must provide written informed consent/assent. For minor patients (ages 12 to 17 years, or as applicable per local regulations), the written ICF must be signed and dated by the parent/legal guardian and the written assent form must be signed and dated by the patient (if applicable). Note: Age requirements are as specified by local regulations.
5. Outpatient >= 12 years of age on the date of consent/assent. In countries where the local regulations permit enrollment of adult patients only, patients must be 18 years of age and older.
6. Asthma diagnosis: The patient has a diagnosis of asthma as defined by the National Institutes of Health (NIH). The asthma diagnosis has been present for a minimum of 3 months and has been stable (defined as no exacerbations and no changes in asthma medication) for at least 30 days.
7. The patient is able to perform acceptable and repeatable spirometry.
8. The patient is able to perform peak expiratory flow (PEF) with a handheld peak flow meter.
9. The patient is able to use a MDI device without a spacer device and a MDPI device.
10. The patient is able to withhold (as judged by the investigator) his or her regimen of ICS or study drug, and rescue medication for at least 6 hours before the SV and before all treatment visits.
11. The patient/parent/legal guardian/caregiver is capable of understanding the requirements, risks, and benefits of study participation, and, as judged by the investigator, capable of giving informed consent/assent and being compliant with all study requirements.
12. SABAs: All patients must be able to replace their current SABA with albuterol/salbutamol HFA MDI inhalation aerosol for the duration of the study.
13. Female patients may not be pregnant, breastfeeding, or attempting to become pregnant.

    * other criteria may apply, please contact the investigator for more information

Exclusion Criteria:

1. A history of a life-threatening asthma exacerbation (an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest, or hypoxic seizures).
2. The patient is pregnant or lactating, or plans to become pregnant during the study period or for 30 days after the study.
3. The patient has participated as a randomized patient in any investigational drug study within 30 days of the SV.
4. The patient has previously participated as a randomized patient in a study of Fp MDPI or FS MDPI.
5. The patient has a known hypersensitivity to any corticosteroid, salmeterol, or any of the excipients in the study drug or rescue medication formulation (ie, lactose).
6. The patient has been treated with any known strong cytochrome P450 (CYP) 3A4 inhibitors (eg, azole antifungals, ritonavir, or clarithromycin) within 30 days before the SV.
7. The patient has been treated with any of the prohibited medications during the prescribed (per protocol) washout periods before the SV.
8. The patient currently smokes or has a smoking history of 10 pack years or more (a pack year is defined as smoking 1 pack of cigarettes/day for 1 year). The patient must not have used tobacco products within the past year (eg, cigarettes, cigars, chewing tobacco, or pipe tobacco).
9. The patient has a culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus, or middle ear that has not resolved at least 2 weeks before the SV.
10. The patient has a history of alcohol or drug abuse within 2 years preceding the SV.
11. The patient has had an asthma exacerbation requiring systemic corticosteroids within 30 days before the SV, or has had any hospitalization for asthma within 2 months before the SV.
12. Initiation or dose escalation of immunotherapy (administered by any route) is planned during the study period. However, patients on stable immunotherapy may be considered for inclusion.
13. The patient has used immunosuppressive medications within 4 weeks before the SV.
14. The patient is unable to tolerate or unwilling to comply with the appropriate washout periods and withholding of all applicable medications.
15. The patient has untreated oral candidiasis at the SV. Patients with clinical visual evidence of oral candidiasis who agree to receive treatment and comply with appropriate medical monitoring may enter the study.
16. The patient has a history of a positive test for human immunodeficiency virus (HIV), active hepatitis B virus, or hepatitis C infection.
17. The patient is either an employee or an immediate relative of an employee of the clinical investigational center.
18. A member of the patient's household is participating in the study at the same time. However, after the enrolled patient completes or discontinues participation in the study, another patient from the same household may be screened.
19. The patient has a disease/condition that in the medical judgment of the investigator would put the safety of the patient at risk through participation or that could affect the efficacy or safety analysis if the disease/condition worsened during the study.

    * other criteria may apply, please contact the investigator for more information

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 787 (Actual)
Dates: Start 2014-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (140):
- United States (76):
  - Teva Investigational Site 12397, Birmingham, Alabama
  - Teva Investigational Site 12375, Glendale, Arizona
  - Teva Investigational Site 12395, Cypress, California
  - Teva Investigational Site 12476, Encinitas, California
  - Teva Investigational Site 12586, Fountain Valley, California
  - Teva Investigational Site 12591, Fresno, California
  - Teva Investigational Site 12372, Huntington Beach, California
  - Teva Investigational Site 12365, Los Angeles, California
  - Teva Investigational Site 12381, Los Angeles, California
  - Teva Investigational Site 12401, Los Angeles, California
  - Teva Investigational Site 12394, Mission Viejo, California
  - Teva Investigational Site 12490, Rancho Mirage, California
  - Teva Investigational Site 12393, Riverside, California
  - Teva Investigational Site 12366, Rolling Hills Estates, California
  - Teva Investigational Site 12383, San Diego, California
  - Teva Investigational Site 12370, San Jose, California
  - Teva Investigational Site 12371, Stockton, California
  - Teva Investigational Site 12579, Upland, California
  - Teva Investigational Site 12379, Centennial, Colorado
  - Teva Investigational Site 12386, Centennial, Colorado
  - Teva Investigational Site 12596, Colorado Springs, Colorado
  - Teva Investigational Site 12584, Longmont, Colorado
  - Teva Investigational Site 12484, Waterbury, Connecticut
  - Teva Investigational Site 12590, Waterbury, Connecticut
  - Teva Investigational Site 12493, Clearwater, Florida
  - Teva Investigational Site 12992, Largo, Florida
  - Teva Investigational Site 12376, Miami, Florida
  - Teva Investigational Site 12390, Miami, Florida
  - Teva Investigational Site 12583, Orlando, Florida
  - Teva Investigational Site 12481, Tallahassee, Florida
  - Teva Investigational Site 12491, Winter Park, Florida
  - Teva Investigational Site 12997, Decatur, Georgia
  - Teva Investigational Site 12392, Savannah, Georgia
  - Teva Investigational Site 12592, Shiloh, Illinois
  - Teva Investigational Site 12483, Lenexa, Kansas
  - Teva Investigational Site 12399, Baltimore, Maryland
  - Teva Investigational Site 12391, Bethesda, Maryland
  - Teva Investigational Site 12589, Columbia, Maryland
  - Teva Investigational Site 12369, Rockville, Maryland
  - Teva Investigational Site 12396, Fall River, Massachusetts
  - Teva Investigational Site 12384, North Dartmouth, Massachusetts
  - Teva Investigational Site 12585, North Dartmouth, Massachusetts
  - Teva Investigational Site 12588, Ypsilanti, Michigan
  - Teva Investigational Site 12494, St Louis, Missouri
  - Teva Investigational Site 12595, St Louis, Missouri
  - Teva Investigational Site 12594, Missoula, Montana
  - Teva Investigational Site 12385, Ocean City, New Jersey
  - Teva Investigational Site 12380, Skillman, New Jersey
  - Teva Investigational Site 12587, Brooklyn, New York
  - Teva Investigational Site 12485, Rockville Centre, New York
  - Teva Investigational Site 12475, Huntersville, North Carolina
  - Teva Investigational Site 12364, Raleigh, North Carolina
  - Teva Investigational Site 12374, Canton, Ohio
  - Teva Investigational Site 12480, Cincinnati, Ohio
  - Teva Investigational Site 12492, Cincinnati, Ohio
  - Teva Investigational Site 12487, Middleburg Heights, Ohio
  - Teva Investigational Site 12488, Sylvania, Ohio
  - Teva Investigational Site 12377, Edmond, Oklahoma
  - Teva Investigational Site 12368, Medford, Oregon
  - Teva Investigational Site 12382, Portland, Oregon
  - Teva Investigational Site 12400, Pittsburgh, Pennsylvania
  - Teva Investigational Site 12473, Upland, Pennsylvania
  - Teva Investigational Site 12389, Greenville, South Carolina
  - Teva Investigational Site 12580, Mt. Pleasant, South Carolina
  - Teva Investigational Site 12398, Orangeburg, South Carolina
  - Teva Investigational Site 12991, Knoxville, Tennessee
  - Teva Investigational Site 12990, Cypress, Texas
  - Teva Investigational Site 12373, Dallas, Texas
  - Teva Investigational Site 12402, El Paso, Texas
  - Teva Investigational Site 12582, New Braunfels, Texas
  - Teva Investigational Site 12363, San Antonio, Texas
  - Teva Investigational Site 12482, San Antonio, Texas
  - Teva Investigational Site 12477, Waco, Texas
  - Teva Investigational Site 12478, Murray, Utah
  - Teva Investigational Site 12388, South Burlington, Vermont
  - Teva Investigational Site 12378, Milwaukee, Wisconsin
- Canada (3):
  - Teva Investigational Site 11065, Toronto, Ontario
  - Teva Investigational Site 11067, Montreal, Quebec
  - Teva Investigational Site 11068, Vancouver, Quebec
- Czechia (3):
  - Teva Investigational Site 54084, Neratovice
  - Teva Investigational Site 54088, Prague
  - Teva Investigational Site 54087, Rokycany
- Hungary (15):
  - Teva Investigational Site 51134, Budapest
  - Teva Investigational Site 51143, Budapest
  - Teva Investigational Site 51144, Budapest
  - Teva Investigational Site 51140, Debrecen
  - Teva Investigational Site 51142, Deszk
  - Teva Investigational Site 51165, Dombóvár
  - Teva Investigational Site 51145, Kiskunhalas
  - Teva Investigational Site 51141, Miskolc
  - Teva Investigational Site 51133, Mosdós
  - Teva Investigational Site 51136, Nyíregyháza
  - Teva Investigational Site 51139, Nyíregyháza
  - Teva Investigational Site 51163, Sopron
  - Teva Investigational Site 51137, Szeged
  - Teva Investigational Site 51164, Szigetvár
  - Teva Investigational Site 51138, Szombathely
- Poland (22):
  - Teva Investigational Site 53182, Bialystok
  - Teva Investigational Site 53183, Bialystok
  - Teva Investigational Site 53185, Bialystok
  - Teva Investigational Site 53191, Bialystok
  - Teva Investigational Site 53187, Bienkówka
  - Teva Investigational Site 53219, Bydgoszcz
  - Teva Investigational Site 53217, Dębica
  - Teva Investigational Site 53178, Krakow
  - Teva Investigational Site 53180, Krakow
  - Teva Investigational Site 53188, Krakow
  - Teva Investigational Site 53220, Lodz
  - Teva Investigational Site 53235, Lodz
  - Teva Investigational Site 53221, Lódz
  - Teva Investigational Site 53237, Lublin
  - Teva Investigational Site 53194, Poznan
  - Teva Investigational Site 53234, Poznan
  - Teva Investigational Site 53233, Strzelce Opolskie
  - Teva Investigational Site 53179, Tarnów
  - Teva Investigational Site 53218, Tarnów
  - Teva Investigational Site 53193, Warsaw
  - Teva Investigational Site 53181, Wroclaw
  - Teva Investigational Site 53189, Wroclaw
- Russia (10):
  - Teva Investigational Site 50236, Chelyabinsk
  - Teva Investigational Site 50227, Kazan'
  - Teva Investigational Site 50234, Moscow
  - Teva Investigational Site 50238, Moscow
  - Teva Investigational Site 50230, Novosibirsk
  - Teva Investigational Site 50224, Saint Petersburg
  - Teva Investigational Site 50231, Saint Petersburg
  - Teva Investigational Site 50233, Voronezh
  - Teva Investigational Site 50237, Yaroslavl
  - Teva Investigational Site 50226, Yekaterinburg
- South Africa (6):
  - Teva Investigational Site 90002, Cape Town
  - Teva Investigational Site 90008, Cape Town
  - Teva Investigational Site 90005, Centurion
  - Teva Investigational Site 90001, Johannesburg
  - Teva Investigational Site 90003, Middelburg
  - Teva Investigational Site 90007, Pretoria
- Ukraine (5):
  - Teva Investigational Site 58125, Kharkiv
  - Teva Investigational Site 58126, Kharkiv
  - Teva Investigational Site 58127, Kyiv
  - Teva Investigational Site 58128, Kyiv
  - Teva Investigational Site 58129, Vinnytsia

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- [Derived] Raphael G, Yiu G, Sakov A, Liu S, Caracta C. Randomized, double-blind trial evaluating the efficacy and safety of fluticasone propionate and fluticasone propionate/salmeterol delivered via multidose dry powder inhalers in patients with persistent asthma aged 12 years and older. J Asthma. 2018 Jun;55(6):640-650. doi: 10.1080/02770903.2017.1350971. Epub 2017 Aug 31. PMID 28763243
- [Derived] Miller DS, Yiu G, Hellriegel ET, Steinfeld J. Dose-ranging study of salmeterol using a novel fluticasone propionate/salmeterol multidose dry powder inhaler in patients with persistent asthma. Allergy Asthma Proc. 2016 Jul;37(4):291-301. doi: 10.2500/aap.2016.37.3963. Epub 2016 May 27. PMID 27216137

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1363 patients with persistent asthma were screened for enrollment into this study. 787 patients at 129 investigational centers in the US and elsewhere internationally met entry criteria and were considered eligible for enrollment into the study.
Pre-assignment Details: Patients were randomized 1:1:1:1:1 to one of the five treatment arms during the Treatment Period.
Groups:
- Enrolled Patients: During the run-in period (from the screening visit to the randomization visit), all patients replaced their current rescue medication with study-specific rescue medication (albuterol/salbutamol HFA MDI) for use on an as-needed basis for the immediate relief of asthma symptoms throughout the period. All patients discontinued their current ICS or ICS/LABA, and took 1 inhalation twice a day from a single-blinded placebo MDPI device and 1 puff twice a day from open-label QVAR 40 mcg HFA MDI (or equivalent).
- Fp MDPI 100 mcg: Patients took 1 inhalation using a multidose dry powder inhaler (MDPI) twice a day of fluticasone propionate for a total daily dose of 200 mcg for 12 weeks.
  Albuterol/salbutamol hydrofluoroalkane (HFA) metered dose inhaler (MDI) was supplied to participants throughout the study to be used as needed as a rescue medication.
- Fp MDPI 50 mcg: Patients took 1 inhalation using a multidose dry powder inhaler (MDPI) twice a day of fluticasone propionate for a total daily dose of 100 mcg for 12 weeks.
  Albuterol/salbutamol hydrofluoroalkane (HFA) metered dose inhaler (MDI) was supplied to participants throughout the study to be used as needed as a rescue medication.
Period: Run-In Period (Pre-assignment)
Arm/Group | Enrolled Patients | FS MDPI 100 / 12.5 mcg | FS MDPI 50 / 12.5 mcg | Fp MDPI 100 mcg | Fp MDPI 50 mcg | Placebo MDPI
Started | 787 (Enrolled) | 0 | 0 | 0 | 0 | 0
Completed | 647 | 0 | 0 | 0 | 0 | 0
Not Completed | 140 | 0 | 0 | 0 | 0 | 0
Not completed — Randomization criteria not met | 70 | 0 | 0 | 0 | 0 | 0
Not completed — Inclusion criteria not met | 30 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 0 | 0 | 0 | 0 | 0
Not completed — Exclusion criteria met | 11 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 8 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 6 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period
Arm/Group | Enrolled Patients | FS MDPI 100 / 12.5 mcg | FS MDPI 50 / 12.5 mcg | Fp MDPI 100 mcg | Fp MDPI 50 mcg | Placebo MDPI
Started | 0 | 129 (Randomized) | 129 (Randomized) | 130 (Randomized) | 129 (Randomized) | 130 (Randomized)
Completed | 0 | 126 | 121 | 121 | 121 | 113
Not Completed | 0 | 3 | 8 | 9 | 8 | 17
Not completed — Adverse Event | 0 | 0 | 3 | 2 | 1 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 2 | 3 | 2
Not completed — Non-compliance | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Disease progression | 0 | 0 | 0 | 1 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 1 | 4
Not completed — Other | 0 | 3 | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | FS MDPI 100 / 12.5 mcg | FS MDPI 50 / 12.5 mcg | Fp MDPI 100 mcg | Fp MDPI 50 mcg | Placebo MDPI | Total
Number analyzed (Participants) | 129 | 129 | 130 | 129 | 130 | 647
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (17.00) | 41.4 (18.61) | 40.6 (17.16) | 43.3 (17.96) | 40.9 (17.35) | 41.5 (17.60)
Age, Customized [Count of Participants; unit: Participants]
  Adolescents (12-17 years) | 19 | 19 | 18 | 13 | 17 | 86
  Adults (18-64 years) | 100 | 97 | 102 | 93 | 102 | 494
  Adults (65+ years) | 10 | 13 | 10 | 23 | 11 | 67
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 71 | 76 | 75 | 70 | 364
  Male | 57 | 58 | 54 | 54 | 60 | 283
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 105 | 109 | 93 | 107 | 101 | 515
  Black or African American | 20 | 19 | 30 | 18 | 26 | 113
  Asian | 4 | 1 | 4 | 1 | 1 | 11
  American Indian or Alaskan Native | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 1
  Other | 0 | 0 | 2 | 2 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 119 | 121 | 114 | 121 | 122 | 597
  Hispanic or Latino | 10 | 8 | 16 | 8 | 7 | 49
  Unknown | 0 | 0 | 0 | 0 | 1 | 1
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.94 (6.686) | 28.00 (7.166) | 27.63 (6.603) | 27.94 (7.259) | 27.99 (6.849) | 27.90 (6.897)
History of Smoking [Count of Participants; unit: Participants]
  Prior smoker | 18 | 13 | 15 | 14 | 12 | 72
  No tobacco use | 111 | 116 | 115 | 115 | 118 | 575
Previous Asthma Therapy [Count of Participants; unit: Participants]
  Inhaled corticosteroid | 97 | 90 | 83 | 89 | 102 | 461
  Inhaled corticosteroid/long-acting beta2-agonist | 32 | 39 | 47 | 40 | 28 | 186
Forced Expiratory Volume in 1 second (FEV1) [Mean (Standard Deviation); unit: liters] — participants with valid measurements (n=126, 128, 129, 129, 129)
  liters | 2.162 (0.5522) | 2.302 (0.6526) | 2.166 (0.5725) | 2.134 (0.6362) | 2.188 (0.5628) | 2.190 (0.5977)

OUTCOME MEASURES:

1. Primary Outcome: Standardized Baseline-Adjusted Forced Expiratory Volume in 1 Second (FEV1) Area Under the Effect Curve From Time Zero to 12 Hours Postdose (FEV1 AUEC0-12h) at Week 12
Description: A subset of approximately 300 patients who performed postdose serial spirometry is based on sample size calculation. Data from these assessments were used to analyze the primary endpoint of baseline adjusted FEV1 AUEC0-12h at week 12 using the trapezoidal rule based on actual time of measurement. It was standardized by dividing it by the number of hours between the start time of dose administration and the end time of the last nonmissing FEV1 measurement.
  The baseline FEV1 was the average of the 2 predose FEV1 measurements (30 and 10 minutes predose). If 1 of these was missing, the nonmissing value was used; if both were missing, baseline was treated as missing. Baseline-adjusted FEV1 was calculated as postdose FEV1 after subtracting the baseline FEV1 value.
Time Frame: Day 1 (predose, baseline), Week 12 and was performed at the following times relative to the administration of study drug (±5 minutes): 15 and 30 minutes and 1, 2, 3, 4, 6, 8, 10, and 12 hours
Population: Full analysis set: a subset of patients who performed postdose serial spirometry at the baseline visit and week 12
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | FS MDPI 100 / 12.5 mcg | FS MDPI 50 / 12.5 mcg | Fp MDPI 100 mcg | Fp MDPI 50 mcg | Placebo MDPI
Number analyzed (Participants) | 61 | 56 | 72 | 63 | 60
liters | 0.408 (0.0465) | 0.399 (0.0479) | 0.254 (0.0434) | 0.268 (0.0457) | 0.074 (0.0487)
Statistical Analysis 1: Comparison: FS MDPI 100 / 12.5 mcg vs Fp MDPI 100 mcg; A fixed-sequence multiple testing procedure was used to control the overall Type I error rate at the 0.05 level (2-sided) for the primary endpoints analyses. Analyses appear in the defined sequence. This is the first in the sequence; Test type: Superiority or Other; p = 0.0076, ANCOVA; Fixed effects of treatment, sex, (pooled) center, previous therapy (ICS or ICS/LABA), and covariates of age and baseline FEV1; LSM difference = 0.154, 95% CI 2-sided [0.041 to 0.267]
Statistical Analysis 2: Comparison: FS MDPI 50 / 12.5 mcg vs Fp MDPI 50 mcg; A fixed-sequence multiple testing procedure was used to control the overall Type I error rate at the 0.05 level (2-sided) for the primary endpoints analyses. Analyses appear in the defined sequence. This is the second in the sequence; Test type: Superiority or Other; p = 0.0322, ANCOVA; [statistical method as in outcome 1, analysis 1]; LSM difference = 0.131, 95% CI 2-sided [0.011 to 0.250]
Statistical Analysis 3: Comparison: FS MDPI 100 / 12.5 mcg vs Placebo MDPI; A fixed-sequence multiple testing procedure was used to control the overall Type I error rate at the 0.05 level (2-sided) for the primary endpoints analyses. Analyses appear in the defined sequence. This is the third in the sequence; Test type: Superiority or Other; p = 0.0000, ANCOVA; [statistical method as in outcome 1, analysis 1]; LSM difference = 0.335, 95% CI 2-sided [0.216 to 0.453]
Statistical Analysis 4: Comparison: FS MDPI 50 / 12.5 mcg vs Placebo MDPI; A fixed-sequence multiple testing procedure was used to control the overall Type I error rate at the 0.05 level (2-sided) for the primary endpoints analyses. Analyses appear in the defined sequence. This is the fourth in the sequence; Test type: Superiority or Other; p = 0.0000, ANCOVA; [statistical method as in outcome 1, analysis 1]; LSM difference = 0.325, 95% CI 2-sided [0.203 to 0.447]

2. Primary Outcome: Change From Baseline in Morning Trough Forced Expiratory Volume in 1 Second (FEV1) at Week 12
Description: Trough FEV1 was a morning spirometry taken predose and pre-rescue bronchodilator. If the patient inadvertently administered asthma medication/study drug at home on the AM of the visit, or if the patient took rescue medication within 6 hours of testing, the visit was rescheduled.
  The baseline for predose FEV1 was defined as the average of the 30-minute and 10-minute predose measurements obtained at the randomization visit (Day 1).
Time Frame: Day 1 (predose, baseline), Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | FS MDPI 100 / 12.5 mcg | FS MDPI 50 / 12.5 mcg | Fp MDPI 100 mcg | Fp MDPI 50 mcg | Placebo MDPI
Number analyzed (Participants) | 126 | 128 | 129 | 128 | 129
liters | 0.315 (0.0352) | 0.319 (0.0350) | 0.204 (0.0340) | 0.172 (0.0347) | 0.053 (0.0350)
Statistical Analysis 1: Comparison: FS MDPI 100 / 12.5 mcg vs Placebo MDPI; A fixed-sequence multiple testing procedure was used to control the overall Type I error rate at the 0.05 level (2-sided) for the primary endpoints analyses. Analyses appear in the defined sequence. This is the fifth in the sequence; Test type: Superiority or Other; p = 0.0000, ANCOVA; Effects due to baseline trough AM FEV1, sex, age, (pooled) center, previous therapy (ICS or ICS/LABA), and treatment; LSM difference = 0.262, 95% CI 2-sided [0.168 to 0.356]
Statistical Analysis 2: Comparison: FS MDPI 50 / 12.5 mcg vs Placebo MDPI; A fixed-sequence multiple testing procedure was used to control the overall Type I error rate at the 0.05 level (2-sided) for the primary endpoints analyses. Analyses appear in the defined sequence. This is the sixth in the sequence; Test type: Superiority or Other; p = 0.0000, ANCOVA; Effects due to baseline trough AM FEV1, sex, age, (pooled) center, previous therapy (ICS or ICS/LABA), and treatment; LSM difference = 0.266, 95% CI 2-sided [0.172 to 0.360]
Statistical Analysis 3: Comparison: Fp MDPI 100 mcg vs Placebo MDPI; A fixed-sequence multiple testing procedure was used to control the overall Type I error rate at the 0.05 level (2-sided) for the primary endpoints analyses. Analyses appear in the defined sequence. This is the seventh in the sequence; Test type: Superiority or Other; p = 0.0017, ANCOVA; Effects due to baseline trough AM FEV1, sex, age, (pooled) center, previous therapy (ICS or ICS/LABA), and treatment; LSM difference = 0.151, 95% CI 2-sided [0.057 to 0.244]
Statistical Analysis 4: Comparison: Fp MDPI 50 mcg vs Placebo MDPI; A fixed-sequence multiple testing procedure was used to control the overall Type I error rate at the 0.05 level (2-sided) for the primary endpoints analyses. Analyses appear in the defined sequence. This is the eighth in the sequence; Test type: Superiority or Other; p = 0.0132, ANCOVA; Effects due to baseline trough AM FEV1, sex, age, (pooled) center, previous therapy (ICS or ICS/LABA), and treatment; LSM difference = 0.119, 95% CI 2-sided [0.025 to 0.212]

3. Secondary Outcome: Change From Baseline in the Weekly Average of the Daily Morning Trough Peak Expiratory Flow (PEF) Over the 12 Week Treatment
Description: Morning PEF tests were performed before administration of study drug or rescue medications (data were excluded if the time of PEF measurement was more than 5 minutes after the dose time). The patient recorded the highest value of 3 measurements obtained in the patient diary. The baseline PEF was the average value of recorded (nonmissing) morning assessments over the 7 days prior to randomization on Day 1. For efficacy analyses of weekly average morning PEF measurements, values were the averages based on available data for that week.
Time Frame: Days -6 to Day 1 (predose), Day 1 (postdose) daily until Week 12
Population: Full analysis set of patients who contributed at least once to the analysis.
Measure: Least Squares Mean (Standard Error); unit: liters/minute
Arm/Group | FS MDPI 100 / 12.5 mcg | FS MDPI 50 / 12.5 mcg | Fp MDPI 100 mcg | Fp MDPI 50 mcg | Placebo MDPI
Number analyzed (Participants) | 125 | 128 | 129 | 128 | 128
liters/minute | 24.415 (3.1530) | 24.864 (3.1182) | 14.517 (3.0778) | 10.609 (3.1176) | 3.591 (3.1474)
Statistical Analysis 1: Comparison: Fp MDPI 100 mcg vs Placebo MDPI; The analysis of change from baseline in weekly average of daily (AM predose and pre-rescue bronchodilator) PEF over the 12-week treatment period was performed using an mixed model for repeated measures (MMRM) with an unstructured covariance matrix and with effects due to baseline weekly average of daily AM PEF, sex, age, (pooled) center, previous therapy (ICS or ICS/LABA), week, treatment, and week-by-treatment interaction; Test type: Superiority or Other; p = 0.0123, mixed model for repeated measures — Significance level of 0.05; LSM difference = 10.926, 95% CI 2-sided [2.380 to 19.471]
Statistical Analysis 2: Comparison: Fp MDPI 50 mcg vs Placebo MDPI; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.1074, mixed model for repeated measures — Significance level of 0.05; LSM difference = 7.018, 95% CI 2-sided [-1.531 to 15.567]
Statistical Analysis 3: Comparison: FS MDPI 100 / 12.5 mcg vs Placebo MDPI; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0000, mixed model for repeated measures — Significance level of 0.05; LSM difference = 20.824, 95% CI 2-sided [12.253 to 29.395]
Statistical Analysis 4: Comparison: FS MDPI 50 / 12.5 mcg vs Placebo MDPI; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0000, mixed model for repeated measures — Significance level of 0.05; LSM difference = 21.273, 95% CI 2-sided [12.728 to 29.818]
Statistical Analysis 5: Comparison: FS MDPI 100 / 12.5 mcg vs Fp MDPI 100 mcg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0233, mixed model for repeated measures — Significance level of 0.05; LSM difference = 9.898, 95% CI 2-sided [1.349 to 18.447]
Statistical Analysis 6: Comparison: FS MDPI 50 / 12.5 mcg vs Fp MDPI 50 mcg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0011, mixed model for repeated measures — Significance level of 0.05; LSM difference = 14.255, 95% CI 2-sided [5.732 to 22.778]
Statistical Analysis 7: Comparison: FS MDPI 50 / 12.5 mcg vs Fp MDPI 100 mcg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0175, mixed model for repeated measures — Significance level of 0.05; LSM difference = 10.347, 95% CI 2-sided [1.822 to 18.872]

4. Secondary Outcome: Change From Baseline in the Weekly Average of the Total Daily Asthma Symptom Score Over the 12-Week Treatment Period
Description: The total daily asthma symptom score is the average of the daytime and nighttime scores as recorded in the patient diary (range 0-9).
  Daytime Symptom Score:
  0=No symptoms
  1. Symptoms for 1 short period
  2. Symptoms for 2+ short periods
  3. Symptoms for most of the day - did not affect normal daily activities
  4. Symptoms for most of the day - did affect normal daily activities
  5. Symptoms so severe that I could not go to work or perform normal daily activities
  Nighttime Symptom Score (determined in the AM):
  0=No symptoms
  1. Symptoms causing me to wake once (or wake early)
  2. Symptoms causing me to wake twice or more (including waking early)
  3. Symptoms causing me to be awake for most of the night
  4. Symptoms so severe that I did not sleep Baseline was the average of recorded scores over the 7 days before randomization. The change from baseline in the weekly average over weeks 1 to 12 was analyzed using an mixed model for repeated measures (MMRM).
Time Frame: Days -6 to Day 1 (predose, baseline) to Week 12
Population: Full analysis set of patients who contributed at least once to the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FS MDPI 100 / 12.5 mcg | FS MDPI 50 / 12.5 mcg | Fp MDPI 100 mcg | Fp MDPI 50 mcg | Placebo MDPI
Number analyzed (Participants) | 125 | 128 | 129 | 128 | 128
units on a scale | -0.364 (0.0318) | -0.329 (0.0314) | -0.300 (0.0308) | -0.278 (0.0314) | -0.135 (0.0318)
Statistical Analysis 1: Comparison: Fp MDPI 100 mcg vs Placebo MDPI; The change from baseline in the weekly average of the total daily asthma symptom scores over weeks 1 to 12 was analyzed using an MMRM with an unstructured covariance matrix and with effects due to baseline score, sex, age, (pooled) center, previous therapy (ICS or ICS/LABA), week, treatment, and week-by-treatment interaction; Test type: Superiority or Other; p = 0.0002, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.165, 95% CI 2-sided [-0.251 to -0.080]
Statistical Analysis 2: Comparison: Fp MDPI 50 mcg vs Placebo MDPI; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0010, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.143, 95% CI 2-sided [-0.229 to -0.058]
Statistical Analysis 3: Comparison: FS MDPI 100 / 12.5 mcg vs Placebo MDPI; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0000, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.230, 95% CI 2-sided [-0.315 to -0.144]
Statistical Analysis 4: Comparison: FS MDPI 50 / 12.5 mcg vs Placebo MDPI; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0000, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.194, 95% CI 2-sided [-0.279 to -0.109]
Statistical Analysis 5: Comparison: FS MDPI 100 / 12.5 mcg vs Fp MDPI 100 mcg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.1381, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.064, 95% CI 2-sided [-0.150 to 0.021]
Statistical Analysis 6: Comparison: FS MDPI 50 / 12.5 mcg vs Fp MDPI 50 mcg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.2438, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.051, 95% CI 2-sided [-0.136 to 0.035]
Statistical Analysis 7: Comparison: FS MDPI 50 / 12.5 mcg vs Fp MDPI 100 mcg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.5095, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.029, 95% CI 2-sided [-0.114 to 0.057]

5. Secondary Outcome: Change From Baseline in the Weekly Average of the Total Daily (24-hour) Use of Albuterol/Salbutamol Inhalation Aerosol Over the 12-Week Treatment Period
Description: Patients recorded the number of inhalations of rescue medication (albuterol/salbutamol HFA MDI) each AM and PM in the diary. The average number of daily inhalations over the 7 days before the randomization visit was the baseline value. The weekly average was based on the available data for the 7 days before each analysis week. The change from baseline in the weekly average of total daily (24-hour) use of albuterol/ salbutamol inhalation aerosol (number of inhalations) over weeks 1 to 12 was analyzed using a mixed model for repeated measures.
Time Frame: Days -6 to Day 1 (predose, baseline), up to week 12
Population: FAS of patients who contributed at least once to the analysis
Measure: Least Squares Mean (Standard Error); unit: puffs
Arm/Group | FS MDPI 100 / 12.5 mcg | FS MDPI 50 / 12.5 mcg | Fp MDPI 100 mcg | Fp MDPI 50 mcg | Placebo MDPI
Number analyzed (Participants) | 126 | 128 | 129 | 128 | 129
puffs | -0.677 (0.0937) | -0.706 (0.0930) | -0.466 (0.0915) | -0.467 (0.0928) | -0.003 (0.0937)
Statistical Analysis 1: Comparison: Fp MDPI 100 mcg vs Placebo MDPI; The change from baseline in the weekly average of total daily (24-hour) use of albuterol/ salbutamol inhalation aerosol (number of inhalations) over weeks 1 to 12 was analyzed using an MMRM with an unstructured covariance matrix and with effects due to baseline value, sex, age, (pooled) center, previous therapy (ICS or ICS/LABA), week, treatment, and week-by-treatment interaction; Test type: Superiority or Other; p = 0.0004, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.463, 95% CI 2-sided [-0.716 to -0.209]
Statistical Analysis 2: Comparison: Fp MDPI 50 mcg vs Placebo MDPI; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0003, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.464, 95% CI 2-sided [-0.718 to -0.211]
Statistical Analysis 3: Comparison: FS MDPI 100 / 12.5 mcg vs Placebo MDPI; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0000, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.675, 95% CI 2-sided [-0.928 to -0.421]
Statistical Analysis 4: Comparison: FS MDPI 50 / 12.5 mcg vs Placebo MDPI; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0000, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.704, 95% CI 2-sided [-0.957 to -0.450]
Statistical Analysis 5: Comparison: FS MDPI 100 / 12.5 mcg vs Fp MDPI 100 mcg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.1014, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.212, 95% CI 2-sided [-0.465 to 0.042]
Statistical Analysis 6: Comparison: FS MDPI 50 / 12.5 mcg vs Fp MDPI 50 mcg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0640, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.239, 95% CI 2-sided [-0.492 to 0.014]
Statistical Analysis 7: Comparison: FS MDPI 50 / 12.5 mcg vs Fp MDPI 100 mcg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0626, mixed model for repeated measures — Significance level of 0.05; LSM difference = -0.241, 95% CI 2-sided [-0.494 to 0.013]

6. Secondary Outcome: Kaplan-Meier Estimate of Probability of Remaining in Study At Week 12
Description: The analysis of probability of remaining in the study at Week 12 used the time to patient withdrawal for worsening asthma, defined as the number of days elapsed from the date of randomization to the date of withdrawal due to worsening asthma. Patients who were lost to follow-up, who had not withdrawn due to worsening asthma by week 12, or who had withdrawn due to reasons other than worsening asthma were right-censored at the date of last assessment.
Time Frame: up to Week 12 of the Treatment Period
Population: FAS
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | FS MDPI 100 / 12.5 mcg | FS MDPI 50 / 12.5 mcg | Fp MDPI 100 mcg | Fp MDPI 50 mcg | Placebo MDPI
Number analyzed (Participants) | 126 | 128 | 129 | 128 | 129
probability | 1.0000 [1.000 to 1.000] | 0.9917 [0.942 to 0.999] | 0.9919 [0.944 to 0.999] | 0.9919 [0.944 to 0.999] | 0.9681 [0.917 to 0.988]
Statistical Analysis 1: Comparison: Fp MDPI 100 mcg vs Placebo MDPI; Test type: Superiority or Other; p = 0.1679, Log Rank — Significance level of 0.05
Statistical Analysis 2: Comparison: Fp MDPI 50 mcg vs Placebo MDPI; Test type: Superiority or Other; p = 0.1701, Log Rank — Significance level of 0.05
Statistical Analysis 3: Comparison: FS MDPI 100 / 12.5 mcg vs Placebo MDPI; Test type: Superiority or Other; p = 0.0437, Log Rank — Significance level of 0.05
Statistical Analysis 4: Comparison: FS MDPI 50 / 12.5 mcg vs Placebo MDPI; Test type: Superiority or Other; p = 0.1718, Log Rank — Significance level of 0.05
Statistical Analysis 5: Comparison: FS MDPI 100 / 12.5 mcg vs Fp MDPI 100 mcg; Test type: Superiority or Other; p = 0.3134, Log Rank — Significance level of 0.05
Statistical Analysis 6: Comparison: FS MDPI 50 / 12.5 mcg vs Fp MDPI 50 mcg; Test type: Superiority or Other; p = 0.9930, Log Rank — Significance level of 0.05
Statistical Analysis 7: Comparison: FS MDPI 50 / 12.5 mcg vs Fp MDPI 100 mcg; Test type: Superiority or Other; p = 0.9999, Log Rank — Significance level of 0.05

7. Secondary Outcome: Change From Baseline in the Asthma Quality of Life Questionnaire With Standardized Activities (AQLQ(S)) Score at Endpoint for Patients >=18 Years Old
Description: The AQLQ(S) (September 2010 version; patients aged ≥18 years) was self-administered by the patients at the investigational center at the randomization visit and at Week 12 or end of trial. The questionnaire is a tool to measure the impact of asthma on a patient's quality of life (physical, emotional, social, and occupational) with a recall period of 2 weeks. The AQLQ(S) was administered only to patients 18 years and older. The 32 individual questions in the AQLQ were equally weighted. The overall AQLQ score was the mean of the responses to each of the 32 questions, and ranged from 1 to 7. A score of 7.0 indicated that the patient had no impairments due to asthma and a score of 1.0 indicated severe impairment.
  Positive change from baseline scores indicate improved quality of life.
Time Frame: Day 1 (predose, baseline), end of trial (up to week 12)
Population: FAS patients who contributed at least once to analysis and were >= 18 years old
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FS MDPI 100 / 12.5 mcg | FS MDPI 50 / 12.5 mcg | Fp MDPI 100 mcg | Fp MDPI 50 mcg | Placebo MDPI
Number analyzed (Participants) | 109 | 102 | 103 | 108 | 97
units on a scale | 0.808 (0.0728) | 0.565 (0.0752) | 0.636 (0.0736) | 0.588 (0.0733) | 0.335 (0.0777)
Statistical Analysis 1: Comparison: Fp MDPI 100 mcg vs Placebo MDPI; The change from baseline in AQLQ(S) score (patients ≥18 years of age) at endpoint (ie, last postbaseline observation) was analyzed using an ANCOVA model with effects due to baseline AQLQ(S) score, sex, age, (pooled) center, previous therapy (ICS or ICS/LABA), and treatment, imputing missing data via last observation carried forward (LOCF); Test type: Superiority or Other; p = 0.0044, ANCOVA — Significance level of 0.05; LSM difference = 0.301, 95% CI 2-sided [0.094 to 0.508]
Statistical Analysis 2: Comparison: Fp MDPI 50 mcg vs Placebo MDPI; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.0155, ANCOVA — Significance level of 0.05; LSM difference = 0.253, 95% CI 2-sided [0.048 to 0.458]
Statistical Analysis 3: Comparison: FS MDPI 100 / 12.5 mcg vs Placebo MDPI; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.0000, ANCOVA — Significance level of 0.05; LSM difference = 0.473, 95% CI 2-sided [0.270 to 0.676]
Statistical Analysis 4: Comparison: FS MDPI 50 / 12.5 mcg vs Placebo MDPI; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.0293, ANCOVA — Significance level of 0.05; LSM difference = 0.230, 95% CI 2-sided [0.023 to 0.437]
Statistical Analysis 5: Comparison: FS MDPI 100 / 12.5 mcg vs Fp MDPI 100 mcg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.0913, ANCOVA — Significance level of 0.05; LSM difference = 0.172, 95% CI 2-sided [-0.028 to 0.372]
Statistical Analysis 6: Comparison: FS MDPI 50 / 12.5 mcg vs Fp MDPI 50 mcg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.8216, ANCOVA — Significance level of 0.05; LSM difference = -0.023, 95% CI 2-sided [-0.223 to 0.177]
Statistical Analysis 7: Comparison: FS MDPI 50 / 12.5 mcg vs Fp MDPI 100 mcg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.4934, ANCOVA — Significance level of 0.05; LSM difference = -0.071, 95% CI 2-sided [-0.275 to 0.133]

8. Secondary Outcome: Kaplan-Meier Estimates for Time to 15% and 12% Improvement From Baseline in FEV1 Postdose on Day 1
Description: A subset of approximately 300 patients who performed postdose serial spirometry is based on sample size calculation. Baseline FEV1 was the average of 2 FEV1 measurements (30 and 10 minutes predose) on Day 1. If one of these was missing, the other measurement was used as baseline value. If both were missing, baseline was treated as missing. Time to target improvement (15% or 12%) was defined as the time elapsed from the time of first dose to the first time the target improvement in FEV1 was achieved. If an exact target increase was not achieved at a measured timepoint, then the time was estimated by linear interpolation between the timepoint when target was reached and the timepoint immediately before. Patients who did not achieve the target improvement were censored at the time of last serial spirometry assessment.
  Values of 9999 indicate the values could not be estimated which happened when the estimated probability of not achieving target is more than 50%.
Time Frame: Day 1 of the Treatment Period (predose and postdose)
Population: Full analysis set: a subset of patients who performed postdose serial spirometry on Day 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | FS MDPI 100 / 12.5 mcg | FS MDPI 50 / 12.5 mcg | Fp MDPI 100 mcg | Fp MDPI 50 mcg | Placebo MDPI
Number analyzed (Participants) | 61 | 56 | 72 | 63 | 60
hours
  15% improvement | 4.3 [1.070 to NA] — values could not be estimated which happened when the estimated probability of not achieving target is more than 50%. | 1.3 [0.600 to 2.750] | NA [10.190 to NA] — values could not be estimated which happened when the estimated probability of not achieving target is more than 50%. | NA [NA to NA] — values could not be estimated which happened when the estimated probability of not achieving target is more than 50%. | NA [NA to NA] — values could not be estimated which happened when the estimated probability of not achieving target is more than 50%.
  12% improvement | 1.0 [0.460 to 3.720] | 0.5 [0.300 to 1.550] | NA [7.370 to NA] — values could not be estimated which happened when the estimated probability of not achieving target is more than 50%. | NA [3.890 to NA] — values could not be estimated which happened when the estimated probability of not achieving target is more than 50%. | NA [7.270 to NA] — values could not be estimated which happened when the estimated probability of not achieving target is more than 50%.

9. Secondary Outcome: Patients With Treatment-Emergent Adverse Experiences (TEAE) During the Treatment Period
Description: An adverse event was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an AE which prevents normal daily activities. Relationship of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 to Week 12 of the Treatment Period
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | FS MDPI 100 / 12.5 mcg | FS MDPI 50 / 12.5 mcg | Fp MDPI 100 mcg | Fp MDPI 50 mcg | Placebo MDPI
Number analyzed (Participants) | 126 | 128 | 129 | 129 | 129
Participants
  >=1 TEAE | 37 | 46 | 40 | 44 | 47
  >=1 severe TEAE | 2 | 0 | 1 | 1 | 0
  >=1 treatment-related TEAE | 4 | 4 | 5 | 7 | 5
  >=1 severe treatment-related TEAE | 0 | 0 | 0 | 0 | 0
  >=1 serious TEAE | 1 | 0 | 1 | 0 | 2
  >=1 TEAE leading to withdrawal | 0 | 3 | 2 | 1 | 6
  >=1 nonserious TEAE | 36 | 46 | 39 | 44 | 45
  >=1 TEAE resulting in death | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 12
Arm/Group | FS MDPI 100 / 12.5 mcg | FS MDPI 50 / 12.5 mcg | Fp MDPI 100 mcg | Fp MDPI 50 mcg | Placebo MDPI
Serious Adverse Events (participants affected / at risk) | 1/126 | 0/128 | 1/129 | 0/129 | 2/129
Other Adverse Events (participants affected / at risk) | 12/126 | 22/128 | 21/129 | 15/129 | 15/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FS MDPI 100 / 12.5 mcg (N=126) | FS MDPI 50 / 12.5 mcg (N=128) | Fp MDPI 100 mcg (N=129) | Fp MDPI 50 mcg (N=129) | Placebo MDPI (N=129)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FS MDPI 100 / 12.5 mcg (N=126) | FS MDPI 50 / 12.5 mcg (N=128) | Fp MDPI 100 mcg (N=129) | Fp MDPI 50 mcg (N=129) | Placebo MDPI (N=129)
Nasopharyngitis (Infections and infestations) | 3 (3) | 11 (11) | 9 (10) | 7 (8) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 6 (6) | 4 (4) | 7 (8) | 6 (6)
Headache (Nervous system disorders) | 7 (10) | 7 (8) | 9 (11) | 2 (4) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.